CLINICAL TRIAL: NCT04564053
Title: A Randomized, Participant and Investigator Blinded, Placebo Controlled, Single Ascending Dose Study Investigating the Safety, Tolerability and Pharmacokinetics of LNA043 in Japanese Participants Wit Osteoarthritis of the Knee
Brief Title: Study of Safety, Tolerability and Pharmacokinetics of LNA043 in Japanese Osteoarthritis Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLNA043A11101
Record Dates: First submitted 2020-09-23; First posted 2020-09-25 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Osteoarthritis; Knee
Keywords: osteoarthritis; knee; cartilage
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Intervention Model Description: This is a non-confirmatory, randomized, participant- and investigator-blinded, placebo-controlled, single ascending dose study.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LNA043 (Experimental): LNA043
  Interventions: Drug: LNA043; Drug: Placebo
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LNA043 — Single intra-articular injection on Day 1
  Arms: LNA043
Drug: Placebo — Single intra-articular injection on Day 1

SUMMARY:
The objective of this study was to determine the safety, tolerability and pharmacokinetics after single ascending dose of LNA043 in Japanese participants with osteoarthritis of the knee.

DETAILED DESCRIPTION:
This was a non-confirmatory, randomized, participant- and investigator-blinded, placebo-controlled, single ascending dose study to investigate the safety, tolerability and PK of LNA043 in Japanese participants with osteoarthritis of the knee. This study consisted of 2 cohorts with a total of 12 participants.

ELIGIBILITY:
Inclusion Criteria:

* Male and female Japanese participants aged 20 to 80 years at screening
* A body mass index (BMI) 16.0 kg/m2 or more but less than 35.0 kg/m2 at screening
* Established diagnosis of primary tibio-femoral osteoarthritis of the target knee by standard American College of Rheumatology (ACR) criteria for at least 6 months prior to screening (clinical and radiological criteria).

Exclusion Criteria:

* Partial or complete joint replacement in the target knee. Planned knee surgery for either knee during the study.
* Arthroscopy of the target knee within 6 months prior to Screening or planned during the study
* Use of electrotherapy, acupuncture, and/or chiropractic treatments for osteoarthritis of the knee within 4 weeks prior to screening
* Malalignment >10° in the target knee (varus/valgus)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | Up to Day 22
  To assess the safety and tolerability of single intra-articular injection of LNA043 in Japanese participants with osteoarthritis of the knee

SECONDARY OUTCOMES:
Area under the serum concentration-time curve of LNA043 from zero to the last measurable concentration | 0 (pre-dose), 0.25, 2, 4, 8, 12, 24, 36, 48, 72, 168 hours post-dose
  To assess systemic PK of LNA043 following single intra-articular injection of LNA043 in Japanese participants with osteoarthritis of the knee
Observed maximum serum concentration of LNA043 | 0 (pre-dose), 0.25, 2, 4, 8, 12, 24, 36, 48, 72, 168 hours post-dose
  To assess systemic PK of LNA043 following single intra-articular injection of LNA043 in Japanese participants with osteoarthritis of the knee
Number of participants with anti-LNA043 antibodies in serum | Day 1 (pre-dose), 4, 8, 15, 22
  To assess systemic immunogenicity of LNA043 (anti-LNA043 antibodies) following single intra-articular injection of LNA043 in Japanese participants with osteoarthritis of the knee

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Japan (2):
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
  - Novartis Investigative Site, Osaka

IPD SHARING:
Plan to Share IPD: No
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1055